CLINICAL TRIAL: NCT00329381
Title: A26-wk,Randomized,Dble-Blinded,Parallel-Grp,Placebo-Controlled,Multi-Centered Study to Eval.the Effect of Xolair(Omalizumab)on Improving the Tolerability of Spec.Immunotherapy in Patients With at Least Mod. Persistent Allergic Asthma Inadequately Controlled w/Inhaled Corticosteroids
Brief Title: Safety and Efficacy Study of Omalizumab Given Prior to Immunotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Gailen D. Marshall, MD, PhD, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CiGE025AUS23
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2007-01

CONDITIONS: Asthma
Keywords: Allergic; Asthma; Immunotherapy
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo will be compared to Xolair 150-375 mg SQ every 2 or 4 weeks based on body weight and pre treatment IgE level.
  Interventions: Drug: Xolair
- 2 (Experimental): Xolair 150-375 mg SQ every 2 or 4 weeks based on body weight and pre treatment IgE level.
  Interventions: Drug: Xolair

INTERVENTIONS:
Drug: Xolair — Xolair 150-375 mg SQ every 2 or 4 weeks based on body weight and pre treatment IgE level.
  Other Names: Omalizumab (Xolair)
  Arms: 1
Drug: Xolair — Xolair 150-375 mg SQ every 2 or 4 weeks based on body weight and pre treatment IgE level.
  Other Names: Omalizumab (Xolair)
  Arms: 2

SUMMARY:
In patients with at least moderate persistent allergic asthma controlled with inhaled steroids, omalizumab(administered per US product label), when compared to placebo, will provide the participants with significantly improved tolerability of specific allergen immunotherapy (allergy shots) administered per a cluster schedule(rapid build up method).

DETAILED DESCRIPTION:
Omalizumab is an FDA approved anti-IgE drug used to treat allergic asthma. This study is designed to give omalizumab 13 weeks prior to administering rapid build up of specific allergy shot, with an overlap of omalizumab and cluster therapy for 3 weeks. The cluster therapy will take 4 week to complete with maintenance dosage lasting an additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis and history of moderate persistent allergic asthma
* body weight >/= 20kg and </= 150kg
* Total serum IgE >/= 30 and </= 700IU/mL
* on a stable asthma treatment including corticosteroids for the preceding 4 weeks
* non smoker for at least 1 year prior to visit 1

Exclusion Criteria:

* patients with severe asthma
* history of immunotherapy to any allergen within the past 3 years
* history of anaphylactic allergic reaction
* upper respiratory tract infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of omalizumab on systemic allergic reactions to specific immunotherapy (SIT) in patients with persistent allergic asthma who require treatment with inhaled steroids | 2005-2007

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D. Marshall, MD/PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States